CLINICAL TRIAL: NCT06234605
Title: A Phase 1b, Open-Label, Safety, Tolerability, and Efficacy Study of HC- 7366 in Combination With Belzutifan (WELIREG™) in Patients With Locally Advanced or Metastatic Renal Cell Carcinoma
Brief Title: A Study of HC-7366 in Combination With Belzutifan (WELIREG™) in Patients With Renal Cell Carcinoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: HiberCell, Inc. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HC366-RCC2311; MK-6482-030 (Other: Merck Sharp & Dohme LLC)
Record Dates: First submitted 2024-01-09; First posted 2024-01-31 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Renal Cell Carcinoma
Keywords: ccRCC; belzutifan; kidney cancer; metastatic; locally advanced; HC-7366; WELIREG™
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms; Neoplasm Metastasis | interventions — belzutifan

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Monotherapy (Experimental): Participants will receive HC-7366 monotherapy [dose to be determined] daily
  Interventions: Drug: HC-7366
- Combination (Experimental): Participants will receive HC-7366 monotherapy [dose to be determined] in combination with belzutifan [120 mg] daily
  Interventions: Drug: HC-7366; Drug: Belzutifan

INTERVENTIONS:
Drug: HC-7366 — HC-7366 is a novel, orally administered, highly selective and potent general control nonderepressible 2 (GCN2) kinase activator.
Drug: Belzutifan — Belzutifan is a potent and selective HIF-2α inhibitor
  Other Names: WELIREG™; MK-6482
  Arms: Combination

SUMMARY:
This is a Phase 1b, open-label, multicenter, safety, tolerability and efficacy study of HC-7366 in combination with belzutifan (WELIREG™). This is a multipart study that consists of a HC-7366 monotherapy cohort, a combination dose escalation, and a combination dose expansion. Approximately 80 patients will be enrolled in this study (up to 20 patients will be enrolled into the HC-7366 monotherapy cohort, up to 30 patients into the combination dose escalation, and up to 30 patients into the combination dose expansion). The primary purpose of this study is to determine the maximum tolerated dose of HC-7366 in combination with belzutifan in patients with locally advanced (inoperable) or metastatic RCC with predominantly clear cell histology, irrespective of VHL gene mutation status.

ELIGIBILITY:
Inclusion Criteria:

* Has diagnosis of locally advanced (inoperable) or metastatic RCC with a predominant clear cell component
* Be age 18 years or older (male or female) at the time of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-04-29 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Determination of MTD and RP2D (combination cohorts only) | 30 months
  To identify the maximum tolerated dose (MTD) and/ or recommended Phase 2 dose (RP2D), and evaluate the safety, tolerability and dose-limiting toxicities (DLTs) of HC-7366 in combination with belzutifan in patients with locally advanced (inoperable) or metastatic RCC with predominantly clear cell histology irrespective of VHL gene mutation status

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - University of Arizona Cancer Center, Tucson, Arizona
  - University of California San Diego Moores Cancer Center, La Jolla, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Rocky Mountain Cancer Centers, LLP, Lone Tree, Colorado
  - Yale - New Haven Hospital, New Haven, Connecticut
  - HealthPartners Cancer Research Center, Saint Paul, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Providence Cancer Institute, Portland, Oregon
  - SCRI Oncology Partners, Nashville, Tennessee
  - Texas Oncology, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University Medical Center & Texas Tech Health Science Center, Lubbock, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Swedish Medical Center, Seattle, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - University of Wisconsin - Carbone Cancer Center, Madison, Wisconsin